CLINICAL TRIAL: NCT06058988
Title: Window of Opportunity Assessment of [Fam-]Trastuzumab DERuxtecan-nxki (T-DXd) Brain Tumor Penetration and Efficacy (WOnDER-BT)
Brief Title: Trastuzumab Deruxtecan (T-DXd) for People With Brain Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-208
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Brain Cancer; Glioblastoma; Metastatic Cancer; Leptomeningeal Metastasis; Recurrent Glioblastoma
Keywords: Brain Cancer; Glioblastoma; Metastatic Cancer; Leptomeningeal Metastasis; Recurrent Glioblastoma; Trastuzumab Deruxtecan; T-DXd; 22-208; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma; Neoplasm Metastasis; Meningeal Carcinomatosis | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Participants with Her2-expressing or solid tumors with activating ERBB2 mutations with 1 or more CNS metastases requiring neurosurgical resection/biopsy with no prior T-DXd
  Interventions: Drug: Trastuzumab deruxtecan
- Cohort B (Experimental): Participants with Her2-expressing or solid tumors with activating ERBB2 mutations with 1 or more CNS metastases requiring neurosurgical resection/biopsy with no prior T-DXd and prior T-DXd exposure and with documented radiological CNS progression while on T-DXd, requiring neurosurgical resection/biopsy of 1 or more recurrent metastases, with continuation of T-DXd until prior to surgery
  Interventions: Drug: Trastuzumab deruxtecan
- Cohort C (Experimental): Participants with recurrent glioblastoma requiring neurosurgical resection/biopsy
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — All participants will receive T-DXd prior to indicated brain tumor resection/biopsy
  Other Names: T-DXd

SUMMARY:
The purpose of this study is to find out how much tratuzumab deruxtecan (T-DXd) can penetrate the tumor when injected into the body, and whether T-DXd may be an effective treatment for brain cancers that express the HER2 protein.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age with one or more brain tumors planned for neurosurgical resection/biopsy
* Pathologically-documented glioblastoma; or
* Metastatic cancer that:

  o Has a history of Her2 expression or activating Her2-mutation
* Her2+ defined as 3+ on IHC
* Her2-low defined as IHC1+ or 2+ and ISH- according to ASCO-CAP 2018 Her2 testing guidelines52
* Her2 mutations must be described to be activating, occur at a known hotspot (e.g. exon 20 insertions, S310, G660, R678, L755, D769, L777), or involve the transmembrane, juxtamembrane or tyrosine kinase domains
* Other untreated brain tumors (and prior radiation, including whole-brain and/or stereotactic radiation) are allowed
* Patients with concomitant leptomeningeal metastasis are eligible provided they have parenchymal brain neoplastic disease requiring resection/biopsy
* Prior treatments:

  * Cohort A: Brain parenchymal metastases in patients with Her2-expressing/ERBB2- activating-mutant cancer with no prior T-DXd exposure (T-DXd naïve)
  * Cohort B: Brain parenchymal metastases in patients with Her2-expressing/ERBB2- activating-mutant cancer with prior T-DXd exposure
  * Cohort C: Recurrent glioblastoma
  * For all cohorts: no limit on prior CNS radiation or systemic therapy, including Her2- targeting antibody therapy (including trastuzumab, pertuzumab, trastuzumab emtansine)
* KPS ≥ 60 Or ECOG < 2
* Life expectancy >12 weeks
* Left ventricular ejection fraction ≥50%
* Adequate bone marrow, renal, hepatic, and coagulation parameters (obtained ≤7 days prior to the first day of study treatment):

  * Absolute neutrophil count (ANC) ≥1.5 × 103/μL (granulocyte-colony stimulating factor administration is not allowed within 1 week prior to C1D1)
  * Platelet count ≥10.0x104/μL. Note: Participants requiring ongoing transfusions or growth factor support to maintain platelet count ≥10.0x104/μL are not eligible. (Platelet transfusion is not allowed within 1 week prior to C1D1)
  * Hemoglobin ≥ 8.0 g/dL. Note: Participants requiring ongoing transfusions or growth factor support to maintain hemoglobin ≥8.0 g/dL are not eligible (> 8 g/dL in gastric cancer / gastroesophageal cancer indications). (Red blood cell transfusion is not allowed within 1 week prior to C1D1)
  * Serum albumin ≥ 2.5 g/dL
  * Creatinine clearance ≥30 mL/min, as calculated using the Cockcroft-Gault equation
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 × upper limit of normal (ULN) (<5x ULN in participants with liver metastases)
  * Total bilirubin ≤1.5 × ULN) if no liver metastases or <3 × ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastases at baseline
  * International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤1.0xULN unless on medication known to reversibly alter INR and/or aPTT
* Evidence of post-menopausal status or negative serum pregnancy test for females of childbearing potential who are sexually active with a non-sterilized male partner. For women of childbearing potential, a negative result for serum pregnancy test (test must have a sensitivity of at least 25 mIU/mL) must be available within 7 days of the screening visit and urine beta-human chorionic gonadotropin (β-HCG) pregnancy test prior to each administration of T-DXd.
* Women of childbearing potential are defined as those who are not surgically sterile (i.e.

underwent bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy). Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.

* Female patients of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception, presented in Table 1 from the time of screening and must agree to continue using such precautions for 7 months after the last dose of T-DXd. Note: estrogen/progesterone is contraindicated in ER+ breast cancer, and in other cancers could increase the risk of DVT. Female patients must refrain from breastfeeding while on study and for 7 months after the last dose of T-DXd.
* Non-sterilized male patients who are sexually active with a female partner of childbearing potential must use a condom with spermicide from screening to 4 months after the final dose ofT-DXd. Complete heterosexual abstinence for the drug washout period is an acceptable contraceptive method if it is in line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable. It is strongly recommended for the female partners of a male patient to also use ≥1 highly effective method of contraception throughout this period, as described in Table 1. In addition, male patients should refrain from fathering a child, or freezing or donating sperm from the time of enrollment until 4 months after the last dose of T-DXd; sperm preservation should be considered prior to enrollment in this study.
* Female subjects must not donate, or retrieve for their own use, ova from the time of enrollment through at least 7 months after the final study drug administration. Preservation of ova may be considered prior to enrollment in this study.
* Adequate treatment washout period from prior therapies to allow recovery from any prior treatment-related toxicities before enrollment in the judgment of the Investigator.

Table 1: Highly effective methods of contraception (<1% failure rate) Non-Hormonal Methods

* Total heterosexual abstinence (evaluate in relation to the duration of the clinical study and the preferred and usual lifestyle choice of the participant)
* Vasectomised sexual partner (if partner is the sole sexual partner of the trial participant and that the vasectomised partner has received medical assessment of the surgical success)
* Bilateral tubal occlusion
* Intrauterine device (provided coils are copper banded)

Hormonal Methods

* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (noting relevant contraindications in ER+ breast cancer, and risk of DVT in other cancers)
* oral
* intravaginal
* transdermal
* Progestogen-only hormonal contraception associated with inhibition of ovulation
* oral
* injectable
* implantable
* Intrauterine hormone-releasing system (IUS)

Exclusion Criteria:

* Contraindication or history of allergic reaction to T-DXd
* Significant comorbidities as per investigator evaluation
* Inability to comply with protocol and/or unwilling or not available for follow up assessments or any condition which in the investigator's opinion makes the patient unsuitable for study participation
* Ferrous or other contraindication to MR imaging
* History of myocardial infarction within 6 months before enrollment
* History of symptomatic congestive heart failure (New York Heart Association Class II to IV)
* Corrected QT interval (QTc) prolongation to >470 ms (females) or >450 ms (male) based on12-lead electrocardiogram (ECG)
* Subjects with troponin levels above ULN at screening (as defined by the manufacturer), and without any myocardial related symptoms, should have a cardiologic consultation before enrollment to rule out MI
* History of (noninfectious) interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis can not be ruled out by baseline chest CT at Screening.
* Lung criteria:

  1. Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g. pulmonary emboli within three months of the study enrollment, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.)
  2. Any autoimmune, connective tissue or inflammatory disorders (e.g. Rheumatoid arthritis, Sjogren's, sarcoidosis etc.) where there is documented, or a suspicion of pulmonary involvement at the time of screening.
  3. Prior pneumonectomy (complete)
* Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
* Active primary immunodeficiency, known human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Receipt of live, attenuated vaccine (mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first dose of trastuzumab deruxtecan. Note: Patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of T-DXd.
* Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤ 1 or baseline. Note: Subjects may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to >Grade 2 for at least 3 months prior to [randomization/enrollment/Cycle 1 Day 1] and managed with standard of care treatment) that the investigator deems related to previous anticancer therapy, such as:

  1. Chemotherapy-induced neuropathy
  2. Fatigue
  3. Residual toxicities from prior IO treatment: Grade 1 or Grade 2 endocrinopathies which may include:

  i. Hypothyroidism/hyperthyroidism ii. Type 1 diabetes iii. Hyperglycemia iv. Adrenal insufficiency v. Adrenalitis vi. Skin hypopigmentation (vitiligo)
* Known allergy or hypersensitivity to study treatment or any of the study drug excipients. For patients who are allergic to gadolinium-based agents may receive premedication as per institutional protocol or imaged without contrast at the discretion of the Principal Investigator; reactions will be managed per standard institutional protocol
* History of severe hypersensitivity reactions to other monoclonal antibodies
* Pregnant or breastfeeding female patients, or patients who are planning to become pregnant.
* Patients with substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
* Multiple primary malignancies within 3 years, with the exception of:

  1. adequately resected non-melanoma skin cancer
  2. carcinoma in situ of the cervix
  3. Smoldering pre-malignant or malignant conditions with minimal concern for CNS or extracranial progression during treatment such as CLL or MGUS based on the assessment of the treating provider
  4. curatively treated in-situ disease
  5. other solid tumors curatively treated
  6. contralateral breast cancer [patients with metastatic breast cancer].
* A pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or Cell-free and Concentrated Ascites Reinfusion Therapy (CART)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2027-09-22 (Estimated); Study Completion 2027-09-22 (Estimated)

PRIMARY OUTCOMES:
Intraoperative plasma concentrations in brain tumors after T-DXd injections | Up to 24 months
  To evaluate the brain tumor penetration of trastuzumab deruxtecan (T-DXd) and its payload (DXd) in Her2+/Her2-low/Her2-mutant brain metastases and of Her2-expressing glioblastoma. Concentrations will be presented as brain tumor:plasma ratios across brain lesions, using intraoperative plasma concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Moss, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org